CLINICAL TRIAL: NCT00659893
Title: A Multi-center, Open Label, Dose-area Escalation, Cohort Study to Evaluate the Safety and Tolerability of 0.05% PEP005 Topical Gel Applied for Two Consecutive Days to Treatment Area(s) of up to a Total of 100 cm2 in Patients With Actinic Keratoses on the Extensor (Dorsal Aspect) Forearm(s)
Brief Title: Safety and Toleration of PEP005 Topical Gel When Applied to a Treatment Area of up to 100cm2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peplin (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PEP005-022
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2008-11

CONDITIONS: Actinic Keratosis
Keywords: Peplin; PEP005; Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- 1 (Experimental): Cohort 1 One 25 cm2 treatment area; on one arm
  Interventions: Drug: PEP005 Topical gel
- 2 (Experimental): Cohort 2 One 50cm2 contiguous treatment area; on one arm
  Interventions: Drug: PEP005 Topical gel
- 3 (Experimental): Cohort 3 Two 25cm2 treatment areas; one on each arm
  Interventions: Drug: PEP005 Topical gel
- 4 (Experimental): Cohort 4 One 25cm2 treatment area; and one 50cm2 contiguous treatment area; one on each arm
  Interventions: Drug: PEP005 Topical gel
- 5 (Experimental): Cohort 5 One 75cm2 contiguous treatment area; on one arm
  Interventions: Drug: PEP005 Topical gel
- 6 (Experimental): Cohort 6 Two 50cm2 contiguous treatment area; one on each arm
  Interventions: Drug: PEP005 Topical gel
- 7 (Experimental): Cohort 7 One 25cm2 treatment area; and one 75cm2 contiguous treatment area; one on each arm
  Interventions: Drug: PEP005 Topical gel
- 8 (Experimental): Cohort 8 One 100cm2 contiguous treatment area; on one arm
  Interventions: Drug: PEP005 Topical gel

INTERVENTIONS:
Drug: PEP005 Topical gel — 0.05%, two day dose

SUMMARY:
Study Hypothesis: Safety and Tolerability will differ when treating multiple contiguous 25 cm2 treatment areas, as compared to individual 25 cm2 treatment areas.

ELIGIBILITY:
Inclusion Criteria:

* Must be male and at least 18 years of age.
* A 100 cm2 contiguous treatment area on each of the right and left extensor (dorsal aspect) forearms, each containing a minimum of 5 AK lesions.

Exclusion Criteria:

* Cosmetic or therapeutic procedures (e.g., use of liquid nitrogen, surgical excision, curettage, dermabrasion, medium or greater depth chemical peel, laser resurfacing): within 2 weeks and within 2 cm of the selected treatment area(s).
* Treatment with immunomodulators, or interferon/ interferon inducers or systemic medications that suppress the immune system: within 4 weeks.
* Treatment with 5-FU, imiquimod, diclofenac, or photodynamic therapy: within 8 weeks and within 2 cm of the selected treatment area(s).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (incidence of AEs, SAEs and skin responses) | Screening to End of Study (Day 57)

CONTACTS AND LOCATIONS:
Overall Officials: George Schmieder, DO, Principal Investigator — Park Avenue Dermatology; Stephen Shumack, MD, Principal Investigator — St George Dermatology and Skin and Cancer Centre
Locations (13):
- United States (8):
  - Radiant Research, Tucson, Arizona
  - Skin Surgery Medical Group Inc., San Diego, California
  - Park Avenue Dermatology, Orange Park, Florida
  - Advanced Dermatology and Cosmetic Surgery, Ormond Beach, Florida
  - Radiant Research Inc., Pinellas Park, Florida
  - Medaphase Inc, Newnan, Georgia
  - Karen S. Harkaway, MD LLC, Riverside Park, New Jersey
  - J&S Studies, College Station, Texas
- Australia (5):
  - St George Dematology and Skin and Cancer Centre, Kogarah, Sydney, New South Wales
  - South East Dermatology, Belmont Specialist Centre, Carina Heights, Brisbane, Queensland
  - Skin and Cancer Foundation, Carlton, Melbourne, Victoria
  - St John of God Dermatology, Subiaco, Perth, Western Australia
  - Burswood Dermatology, Victoria Park, Perth, Western Australia

REFERENCES:
- [Derived] Anderson L, Jarratt M, Schmieder G, Shumack S, Katsamas J, Welburn P. Tolerability and Pharmacokinetics of Ingenol Mebutate 0.05% Gel Applied to Treatment Areas up to 100cm(2) on the Forearm(s) of Patients with Actinic Keratosis. J Clin Aesthet Dermatol. 2014 Dec;7(12):19-29. PMID 25584134
- See also: Food and Drug Administration — http://www.fda.gov
- See also: Therapeutic Goods Administration — http://www.tga.gov.au/